CLINICAL TRIAL: NCT04582019
Title: A Single-center Randomized, Controlled Study Evaluating Safety and Effectiveness of Ureteral dj Stent With Magnet (Blackstar, Urotech), Stent-related Symptoms and Pain Level After Stent Removal Compared With Conventional Stent Removal With Flexible Cystoscope
Brief Title: Safety and Effectiveness of Ureteral DJ Stent With Magnet (Blackstar, Urotech) Removal Under Ultrasound Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, nariman.gadjiev, Head of endourology department, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/20-н
Record Dates: First submitted 2020-09-25; First posted 2020-10-09 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: * group A - male patients who will undergo ureteral stent placement by conventional polyurethane DJ stent, Fr 6.5. N=30
  * group B - male patients who will undergo ureteral stent placement by polyurethane DJ stent with magnet (Blackstar, Urotech ), Fr 7. N=30
Who Masked: Investigator
Masking Description: Patients are to be assigned a randomization number that will match their treatment. Block randomization using 10 blocks is to be performed by a central randomization organization (www.randomize.net) using a computerized algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with polyurethane DJ stent (Active Comparator): Polyurethane DJ stent, 6Fr. The stent will be removed using flexible cystoscopy.
  Interventions: Device: stent extraction
- Patients with polyurethane DJ stent with magnet (Active Comparator): Polyurethane DJ stent with magnet (Blackstar, Urotech), 7Fr. The stent will be removed under ultrasound control using a magnetic retriever
  Interventions: Device: stent extraction

INTERVENTIONS:
Device: stent extraction — stent extraction using magnetic retriever or flexible cystoscope

SUMMARY:
Evaluation of safety and effectiveness of ureteral DJ stent with magnet (Blackstar, Urotech), severity of stent-association symptoms and pain level syndrome after stent extraction compared with stent extraction by flexible cystoscope

DETAILED DESCRIPTION:
Inclusion Criteria:

* age from 18 to 70 years
* males
* Indications for rigid or flexible URS
* ASA score: 1-3

Exclusion Criteria:

* Active urinary tract infection
* taking alpha-1 adreno and M-cholinoblockers

All patients will be randomized into 2 groups:

* group A - male patients who will undergo ureteral stent placement by conventional polyurethane DJ stent, Fr 6.5. N=30
* group B - male patients who will undergo ureteral stent placement by polyurethane DJ stent with magnet (Blackstar, Urotech ), Fr 7. N=30 Patients are to be assigned a randomization number that will match their treatment. Block randomization using 10 blocks is to be performed by a central randomization organization (www.randomize.net) using a computerized algorithm.

Using the Visual Analog Scale of Pain (VASP) and Ureteric Stent Symptom Questionnaire (USSQ) we are going to assess the pain syndrome and the severity of stent-associated symptoms. The USSQ will be filled twice: 3 days after stent placement and on the day of stent removal, just before the procedure. All stents will be removed 30 days after placement. Also, immediately after stent removal, patients will complete the VASP questionnaire. In the control group, the stent will be removed using flexible cystoscopy. In the experimental group under ultrasound control using a magnetic retriever, with a bladder capacity of at least 150 ml.

Primary assessed outcomes:

1. Age
2. Body mass index
3. Operation side
4. The density of the stone
5. Type of the operation
6. Applying of the ureteral accessing sheath
7. Type of the ureteral stent
8. Troubles with stent placement
9. USSQ (Ureteral stent symptom questionnaire) 3 days after surgery
10. USSQ before stent extraction
11. VASP (Visual Analog Scale Pain) immediately after stent extraction
12. Duration of stent extractiom by magnetic retrieval device
13. Duration of stent extraction by cystoscopy
14. Stent removal success (yes/no)

Secondary assessed outcomes:

1. Assessment of Stone-free status after surgery by performing computed tomography of kidneys and urinary tract without intravenous contrasting 1 month after surgery
2. Stent encrustation

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 70 years
* males
* Indications for rigid or flexible URS
* ASA score: 1-3

Exclusion Criteria:

* Active urinary tract infection
* taking alpha-1 adreno and M-cholinoblockers

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Stent-related symptoms (SRS) | 30 days
  Using USSQ to evaluate the difference of SRS in patients with different types of stent
Body pain | 30 days
  Using VASP to evaluate the pain level in patients with different types of stent extraction

CONTACTS AND LOCATIONS:
Locations (1):
- First Pavlov Saint Petersburg University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No